CLINICAL TRIAL: NCT05740683
Title: Alpha-synuclein Rt-quic and Neurologic Symptoms in Persons With idiOpathic anosMiA
Acronym: AROMA
Status: Recruiting | Type: Observational
Sponsor: Danish Dementia Research Centre (Network)
Collaborators: Danish Reference Center for Prion Diseases, Rigshospitalet (Unknown); Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Rigshospitalet (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-22053428
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Anosmia; Idiopathic Hyposmia; Idiopathic Olfactory Dysfunction
Keywords: RT-QuIC; alpha-synuclein; Idiopathic anosmia; Idiopathic hyposmia; Idiopathic olfactory dysfunction; Prodromal Parkinsons disease; Prodromal dementia with Lewy bodies
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Olfactory mucosa, skin, saliva and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with idiopathic olfactory dysfunction
  Interventions: Diagnostic Test: RT-QuiC
- People without olfactory dysfunction
  Interventions: Diagnostic Test: RT-QuiC

INTERVENTIONS:
Diagnostic Test: RT-QuiC — RT-QuIC measures the ability of aSyn to misfold other aSyn proteins and is an amplification technique.

SUMMARY:
Test of early warning signs and RT-QuIC in patients with idiopathic olfactory dysfunction

DETAILED DESCRIPTION:
Background. The number of persons living with dementia is increasing in Denmark and worldwide because the population is generally growing older. Dementia with Lewy bodies (DLB) is the second most prevalent etiology among the neurodegenerative diseases that give rise to dementia.

DLB is characterized by many prodromal symptoms years before dementia is evident. Currently, little is known about the course of symptoms in the prodromal phase, and furthermore, the diagnosis of DLB can be clinically challenging, especially in the early stages. DLB is like Parkinson's disease (PD), characterized by the accumulation of alpha-synuclein, which misfolds and aggregates within neurons in so-called Lewy Bodies; this assumably drives the neurodegeneration. A novel technique for the measurement of misfolded alpha-synuclein is Real-Time Quaking-Induced Conversion (RT-QuIC), which may be able to support the diagnostic process as well as aid in identifying patients with prodromal DLB. This would enable earlier symptomatic relief and care and potentially promote the search for disease-modifying therapies, which is currently absent.

Objectives. The overarching objective of this project is to identify early clinical warning signs and biomarkers in prodromal DLB.

Method. Study 1: Exploratory cross-sectional case-control study of patients with olfactory dysfunction versus individuals without olfactory dysfunction assessing pathological alpha-synuclein by RT-QuIC and prodromal symptoms of DLB and Parkinson's Disease.

Study 2: Longitudinal follow-up in Danish registries on diagnosing PD and dementia.

ELIGIBILITY:
Inclusion criteria with patients iOD:

* Age 55 -75 years of age
* Slowly progressing and non-fluctuating iOD
* Able to give informed consent and to cooperate as evaluated by the PI

Exclusion criteria with patients iOD:

* Diagnosed with a neurodegenerative disease or major neurological/psychiatric condition.
* Anosmia/hyposmia caused by sino-nasal disease (including chronic rhinitis and allergy), after trauma, infection, congenial, olfactory dysfunction due to surgery, or toxins/drugs affecting the olfactory function.
* Olfactory dysfunction with response to systemic or local corticosteroids if tried
* Severe nasal cavity abnormalities or infections.
* Overt signs of dementia or PD
* Current alcohol or drug abuse
* Terminal illness
* Diagnosed with neurodegenerative disease or major neurological/psychiatric condition.

Inclusion criteria controls:

* Age 55 -75 years of age
* Able to give informed consent
* Able to cooperate as evaluated by the PI

Exclusion criteria controls:

* Olfactory dysfunction on clinical test
* Overt signs of dementia or PD
* Severe nasal cavity abnormalities or infections.
* Current alcohol or drug abuse
* Diagnosed with neurodegenerative disease or major neurological/psychiatric condition.

Ages: 55 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Fifty patients with idiopathic olfactory dysfunction (iOD) will be recruited from an anosmia clinic and community with posters in relevant newspapers and clinics. Also, 50 controls will be recruited from the community with posters in relevant newspapers and clinics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Real-time quaking-induced conversion (RT-QuIC) positive for alpha-synuclein (aSyn) | 24 months
Diagnosis of Parkinson's disease (PD) or dementia | 8 years
  A diagnosis of PD or dementia in national databases.

SECONDARY OUTCOMES:
Smell test | 24 months
  Sniffin Sticks identification test (SIT16)
Smell test | 24 months
  Sniffin Sticks 48 (score 0-48)
Motor function | 24 months
  Movement Disorder's Unified Parkinson's Rating Scale (MDS-UPDRS-III) (score 0-132)
Dysautonomia and non-motor symptoms | 24 months
  Movement Disorder's Unified Parkinson's Rating Scale (MDS-UPDRS-I) (score 0-52)
Subjective motor symptoms | 24 months
  Movement Disorder's Unified Parkinson's Rating Scale (MDS-UPDRS-II) (score 0-52)
Cognition | 24 months
  MoCA, SDMT, Recall test and fluency (Animals/1 min)
Prodromal PD | 24 months
  MDS Prodromal PD probability
REM-sleep | Ever
  REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ) (score 0-13) and REM Sleep Behavior Disorder Single-Question Screen (RBD1Q)
Color vision | Now
  The Farnsworth-Munsell 100 Hue Color Vision test (score 0-1000)
Co-morbidities and medication | 10 years
  Co-morbidities and medication

CONTACTS AND LOCATIONS:
Overall Officials: Kristian S Frederiksen, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Oskar McWilliam, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Steen G Hasselbalch, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Gunhild Waldemar, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Marie Brunn, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Anja H Simmonsen, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region
Locations (2):
- Denmark (2):
  - Danish Dementia Research Centre, Copenhagen
  - Oskar McWilliam, Copenhagen

IPD SHARING:
Plan to Share IPD: No